CLINICAL TRIAL: NCT03899246
Title: Safety and Feasibility of High-Dose Topical Capsaicin for the Treatment of Neuropathic Pain in Pediatric Sickle Cell Disease
Brief Title: Sickle Cell Pain: Intervention With Capsaicin Exposure
Acronym: SPICE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Michigan (Other)
Responsible Party: Principal Investigator, Alexander Glaros, Pediatric Hematology-Oncology Fellow, Children's Hospital of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPICE1.0
Record Dates: First submitted 2019-01-25; First posted 2019-04-02 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Neuropathic Pain; Sickle Cell Disease
Keywords: Capsaicin; Topical Analgesia; Quantitative Sensory Testing; Pain
MeSH Terms: conditions — Neuralgia; Anemia, Sickle Cell; Pain | interventions — Capsaicin

STUDY DESIGN:
Intervention Model Description: Single arm, safety and feasibility trial assessing the suitability of an FDA approved medication for use in children with an off-label condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Capsaicin Arm (Experimental): Single arm to receive eight percent topical capsaicin applied to up to 4 sites of recurrent pain over one hour on an every three month schedule. Participants in this arm will receive pretreatment with topical five percent lidocaine.
  Interventions: Drug: Eight Percent Topical Capsaicin

INTERVENTIONS:
Drug: Eight Percent Topical Capsaicin — See arm description
  Other Names: Qutenza

SUMMARY:
This study evaluates the safety and feasibility of using high dose topical capsaicin patches for the treatment of neuropathic pain in pediatric patients with sickle cell disease, as well as the feasibility of using a number of tests for the evaluation and monitoring of neuropathic pain. The hypothesis, based on evidence obtained from studies in adults with neuropathic pain related to other diseases as well as a single previously published study of capsaicin in pediatric patients, is that capsaicin will be well tolerated in this population. Additionally, it is hypothesized that it is feasible to monitor changes in neuropathic pain via the testing listed below.

DETAILED DESCRIPTION:
Patients with sickle cell disease suffer debilitating painful episodes, as well as chronic, often daily, pain that are commonly treated with non-steroidal anti-inflammatory drugs, opioids, and other non-pharmacologic supportive measures. Neuropathic pain has been shown to be present in these patients, with frequency increasing with age. It is believed, based on knowledge of neuropathic pain related to other conditions and from the small number of studies in sickle cell patients, to result from repeated vaso-occlusive pain episodes that prime central and peripheral pain sensing pathways in a maladaptive manner, leading to hyper-sensitization. Very few studies to date have evaluated therapies specifically targeting this aspect of the pain experienced by patients with sickle cell disease.

This is a pilot study for a future longitudinal study of neuropathic pain in pediatric patients with sickle cell disease. The first aim of this pilot study is to establish the safety of treating participants with sickle cell disease aged fourteen to twenty-one with eight percent topical capsaicin patches on an every three-month dosing schedule as recommended by the manufacturer. This will be a single-arm safety study. Presence of neuropathic pain will be determined by day zero evaluation via the testing shown in the outcome measures below. Topical medication will be administered over one hour, every three months, for six months (total of three applications), to sites of recurrent vaso-occlusive pain, according to the package insert administration guidelines. Subjective and objective evaluations of pain and inflammation including questionnaires, blood tests, and quantitative sensory testing will be carried out every six weeks throughout the study period until twelve weeks after the final capsaicin application. Additionally, participants will record daily pain and medication use in a mobile app. Safety will be established by there being no grade three or four adverse events according to CTCAE definitions. Grade two adverse events will be evaluated on a case by case basis throughout the duration of the study. Feasibility of monitoring neuropathic pain with the aforementioned studies will be established by participant compliance with greater than eighty percent of all study activities.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of either Sickle Cell Disease with genotype SS or S Beta-zero, or SC disease.
* Must have recurrent sites of pain, where majority of acute pain episodes are localized
* Subjects are willing and able to comply with scheduled visits, treatment plan, laboratory tests, pain assessments, and other study procedures.
* Subjects who are being treated with hydroxyurea (HU) must have been on a stable dose for at least 8 weeks prior to Visit 1 (Day 0), with the intent of remaining on the same dose of hydroxyurea throughout the clinical trial including the protocol-specified follow-up period unless adjustments are medically necessary due to bone marrow suppression.
* At least 80% compliance (defined as logging pain at least once daily) with mobile application use during 14-day lead in period from time of enrollment to time of first capsaicin application.

Exclusion Criteria:

* Age less than 14 or greater than 21
* History of major surgery within the past 3 months.
* Patients receiving scheduled chronic partial exchange transfusions as part of their sickle cell disease management protocol.
* Concurrently taking another medication used in the treatment of neuropathic pain or with the potential to affect the peripheral nervous system (e.g. gabapentin, anti-epileptics, antidepressants, systemic alpha or beta adrenergic receptor blockers)
* Use of another topical analgesic at home in the treatment of pain episodes such as topical lidocaine, diclofenac, or menthol (must discontinue use at the time of enrollment).
* Recurrent pain secondary to an underlying condition other than vaso-occlusive pain (avascular necrosis, scoliosis, fracture, etc.)
* Patients lacking the mental capacity to assent to the study
* Patients with another chronic inflammatory/immune disorder that could skew the inflammatory markers listed above.
* Pregnant females
* Expectation that the subject will not be able to be followed for the duration of the study
* Active use of illicit drugs and/or alcohol dependence, as determined by the investigator. Opioid use beyond the amount necessary for pain related to the underlying sickle cell disease as determined by the investigator.
* Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator.

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE Criteria | At the end of the 9 month study period all participant information will be reviewed and adverse events assessed.
  Safety will be established by there being no treatment-related adverse events greater than grade 2 using CTCAE definitions of adverse events. Grade 2 CTCAE events will be evaluated on a case by case basis to determine safety of continuing the study. Grade 3 events will result in immediate suspension of study activities until a full analysis of the event in question is completed.
Compliance with Serum Substance P Levels | At the end of the 9 month study period all participant information will be reviewed and compliance with testing assessed.
  Feasibility will be established by participants having greater than 80 percent compliance with all study investigations, including serum substance P levels.
Compliance with Subjective Neuropathic Pain Questionnaire | At the end of the 9 month study period all participant information will be reviewed and compliance with testing assessed.
  Feasibility will be established by participants having greater than 80 percent compliance with all study investigations, including completion of PainDETECT Questionnaire during study visits. The questionnaire is a validated assessment of neuropathic pain. It consists of a series of questions regarding the experience of pain for which the participant will provide an answer ranging from "never" (0 points) to "very strongly" (5 points). Points are added to provide a total score from 0 to 38. A score from 0 to 12 indicates a neuropathic pain component is unlikely, a score of 12 to 18 is equivocal, and a score greater than 18 indicates a neuropathic component is likely.
Compliance with Quantitative Sensory Testing | At the end of the 9 month study period all participant information will be reviewed and compliance with testing assessed.
  Feasibility will be established by participants having greater than 80 percent compliance with all study investigations, including quantitative sensory testing using electronic von frey machine.

SECONDARY OUTCOMES:
Compliance with Mobile App Record Keeping | Duration of study period (9 months). Mobile app recordings can be reviewed in real time and will be recorded on a weekly basis.
  Feasibility, as above, will be established by greater than 80 percent compliance with daily mobile app recordings of pain and home medication use.
Compliance with Blood Draws for Hyperspectral Imaging Analysis for Determining Presence and Improvement of Chronic Neuropathic Pain | Duration of study period (9 months). Will be drawn and processed at 6 week intervals throughout the study period.
  Feasibility will be established by the successful processing of greater than 80 percent of target number of blood samples to be sent for hyperspectral analysis, a novel test capable of detecting chronic pain states, but not yet used in the sickle cell population.
Morphine Equivalents Utilized | Duration of study period (9 months). Will be evaluated at 6 week intervals throughout the study period.
  Will assess changes in pain medication required during the course of the study period based on electronic medical record, participant report, and controlled substance monitoring database.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander K Glaros, MD, Principal Investigator — Children's Hospital of Michigan; Ahmar U Zaidi, MD, Principal Investigator — Children's Hospital of Michigan; Callaghan Michael, MD, Principal Investigator — Children's Hospital of Michigan
Locations (1):
- Children's Hospital of Michigan, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith WR, Bovbjerg VE, Penberthy LT, McClish DK, Levenson JL, Roberts JD, Gil K, Roseff SD, Aisiku IP. Understanding pain and improving management of sickle cell disease: the PiSCES study. J Natl Med Assoc. 2005 Feb;97(2):183-93. PMID 15712781
- [Background] Franck LS, Treadwell M, Jacob E, Vichinsky E. Assessment of sickle cell pain in children and young adults using the adolescent pediatric pain tool. J Pain Symptom Manage. 2002 Feb;23(2):114-20. doi: 10.1016/s0885-3924(01)00407-9. PMID 11844631
- [Background] Brandow AM, Farley RA, Panepinto JA. Neuropathic pain in patients with sickle cell disease. Pediatr Blood Cancer. 2014 Mar;61(3):512-7. doi: 10.1002/pbc.24838. Epub 2013 Oct 26. PMID 24167104
- [Background] Brandow AM, Zappia KJ, Stucky CL. Sickle cell disease: a natural model of acute and chronic pain. Pain. 2017 Apr;158 Suppl 1(Suppl 1):S79-S84. doi: 10.1097/j.pain.0000000000000824. No abstract available. PMID 28221286
- [Background] Antunes FD, Propheta VGS, Vasconcelos HA, Cipolotti R. Neuropathic pain in patients with sickle cell disease: a cross-sectional study assessing teens and young adults. Ann Hematol. 2017 Jul;96(7):1121-1125. doi: 10.1007/s00277-017-2984-z. Epub 2017 Mar 30. PMID 28361297
- [Background] Brandow AM, Farley RA, Panepinto JA. Early insights into the neurobiology of pain in sickle cell disease: A systematic review of the literature. Pediatr Blood Cancer. 2015 Sep;62(9):1501-11. doi: 10.1002/pbc.25574. Epub 2015 May 13. PMID 25976161
- [Background] Kenyon N, Wang L, Spornick N, Khaibullina A, Almeida LE, Cheng Y, Wang J, Guptill V, Finkel JC, Quezado ZM. Sickle cell disease in mice is associated with sensitization of sensory nerve fibers. Exp Biol Med (Maywood). 2015 Jan;240(1):87-98. doi: 10.1177/1535370214544275. Epub 2014 Jul 28. PMID 25070860
- [Background] Garrison SR, Kramer AA, Gerges NZ, Hillery CA, Stucky CL. Sickle cell mice exhibit mechanical allodynia and enhanced responsiveness in light touch cutaneous mechanoreceptors. Mol Pain. 2012 Sep 10;8:62. doi: 10.1186/1744-8069-8-62. PMID 22963123
- [Background] Campbell CM, Moscou-Jackson G, Carroll CP, Kiley K, Haywood C Jr, Lanzkron S, Hand M, Edwards RR, Haythornthwaite JA. An Evaluation of Central Sensitization in Patients With Sickle Cell Disease. J Pain. 2016 May;17(5):617-27. doi: 10.1016/j.jpain.2016.01.475. Epub 2016 Feb 16. PMID 26892240
- [Background] Henrich F, Magerl W, Klein T, Greffrath W, Treede RD. Capsaicin-sensitive C- and A-fibre nociceptors control long-term potentiation-like pain amplification in humans. Brain. 2015 Sep;138(Pt 9):2505-20. doi: 10.1093/brain/awv108. Epub 2015 May 4. PMID 25943423
- [Background] Jara-Oseguera A, Simon SA, Rosenbaum T. TRPV1: on the road to pain relief. Curr Mol Pharmacol. 2008 Nov;1(3):255-69. doi: 10.2174/1874467210801030255. PMID 20021438
- [Background] Jessell TM. Substance P in nociceptive sensory neurons. Ciba Found Symp. 1982;(91):225-48. doi: 10.1002/9780470720738.ch13. PMID 6183072
- [Background] Yaksh TL, Farb DH, Leeman SE, Jessell TM. Intrathecal capsaicin depletes substance P in the rat spinal cord and produces prolonged thermal analgesia. Science. 1979 Oct 26;206(4417):481-3. doi: 10.1126/science.228392.
- [Background] Jessell TM, Iversen LL, Cuello AC. Capsaicin-induced depletion of substance P from primary sensory neurones. Brain Res. 1978 Aug 18;152(1):183-8. doi: 10.1016/0006-8993(78)90146-4. No abstract available. PMID 209869
- [Background] Simone DA, Nolano M, Johnson T, Wendelschafer-Crabb G, Kennedy WR. Intradermal injection of capsaicin in humans produces degeneration and subsequent reinnervation of epidermal nerve fibers: correlation with sensory function. J Neurosci. 1998 Nov 1;18(21):8947-59. doi: 10.1523/JNEUROSCI.18-21-08947.1998. PMID 9787000
- [Background] Nolano M, Simone DA, Wendelschafer-Crabb G, Johnson T, Hazen E, Kennedy WR. Topical capsaicin in humans: parallel loss of epidermal nerve fibers and pain sensation. Pain. 1999 May;81(1-2):135-45. doi: 10.1016/s0304-3959(99)00007-x. PMID 10353501
- [Background] Kennedy WR, Vanhove GF, Lu SP, Tobias J, Bley KR, Walk D, Wendelschafer-Crabb G, Simone DA, Selim MM. A randomized, controlled, open-label study of the long-term effects of NGX-4010, a high-concentration capsaicin patch, on epidermal nerve fiber density and sensory function in healthy volunteers. J Pain. 2010 Jun;11(6):579-87. doi: 10.1016/j.jpain.2009.09.019. Epub 2010 Apr 18. PMID 20400377
- [Background] Burness CB, McCormack PL. Capsaicin 8 % Patch: A Review in Peripheral Neuropathic Pain. Drugs. 2016 Jan;76(1):123-34. doi: 10.1007/s40265-015-0520-9. PMID 26666418
- [Background] Rodriguez-Lopez MJ, Fernandez-Baena M, Barroso A, Yanez-Santos JA. Complex Regional Pain Syndrome in Children: a Multidisciplinary Approach and Invasive Techniques for the Management of Nonresponders. Pain Pract. 2015 Nov;15(8):E81-9. doi: 10.1111/papr.12317. Epub 2015 Jun 11. PMID 26095620
- [Background] Brandow AM, Wandersee NJ, Dasgupta M, Hoffmann RG, Hillery CA, Stucky CL, Panepinto JA. Substance P is increased in patients with sickle cell disease and associated with haemolysis and hydroxycarbamide use. Br J Haematol. 2016 Oct;175(2):237-245. doi: 10.1111/bjh.14300. Epub 2016 Aug 19. PMID 27539682
- [Background] Kuei N, Patel N, Xu H, et al. Characteristics and Potential Biomarkers for Chronic Pain in Patients with Sickle Cell Disease. Blood. 2015;126(23). http://www.bloodjournal.org/content/126/23/986?utm_source=TrendMD&utm_medium=cpc&utm_campaign=Blood_TrendMD_0&sso-checked=true. Accessed July 7, 2018.
- [Background] O'Leary JD, Crawford MW, Odame I, Shorten GD, McGrath PA. Thermal pain and sensory processing in children with sickle cell disease. Clin J Pain. 2014 Mar;30(3):244-50. doi: 10.1097/AJP.0b013e318292a38e. PMID 23629596
- [Background] Brandow AM, Panepinto JA. Clinical Interpretation of Quantitative Sensory Testing as a Measure of Pain Sensitivity in Patients With Sickle Cell Disease. J Pediatr Hematol Oncol. 2016 May;38(4):288-93. doi: 10.1097/MPH.0000000000000532. PMID 26907660
- [Background] Staikopoulos V, Gosnell ME, Anwer AG, Mustafa S, Hutchinson MR, Goldys EM. Hyperspectral imaging of endogenous fluorescent metabolic molecules to identify pain states in central nervous system tissue. In: Hutchinson MR, Goldys EM, eds. Vol 10013. International Society for Optics and Photonics; 2016:1001306. doi:10.1117/12.2243158